CLINICAL TRIAL: NCT01015807
Title: Transversus Abdominis Plane (TAP) Block for Cesarean Section
Acronym: CLOTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Laurent Bollag, Assistant Professor, Department of Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36707
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Hyperalgesia, Secondary
Keywords: postoperative; hyperalgesia; pain; transversus abdominis plane block; TAP block; cesarean section
MeSH Terms: conditions — Hyperalgesia; Pain | interventions — Sodium Chloride; Bupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Sterile Saline used for TAP block = Bupivacaine Placebo + Clonidine Placebo
  Interventions: Drug: Bupivacaine Placebo; Drug: Clonidine Placebo
- TAP (Bupi) (Active Comparator): 2x20mL 0.375% Bupivacaine + 2x1mL of 0.9% NaCl = 150mg Bupivacaine + Clonidine Placebo
  Interventions: Drug: Clonidine Placebo; Drug: Bupivacaine
- Clo-TAP (Bupi + Clon) (Active Comparator): 2x20mL 0.375% Bupivacaine + 2x1mL Clonidine = 150mg Bupivacaine + 150µg Clonidine
  Interventions: Drug: Bupivacaine; Drug: Clonidine

INTERVENTIONS:
Drug: Bupivacaine Placebo — 2 x 20mL 0.9% NaCl
  Other Names: Bupi Placebo; Sodium Chloride
  Arms: Placebo
Drug: Clonidine Placebo — 2 x 1mL 0.9% NaCl
  Other Names: Sodium Chloride
  Arms: Placebo; TAP (Bupi)
Drug: Bupivacaine — 2 x 20mL 0.375% Bupivacaine = 150 mg Bupivacaine
  Other Names: Bupivacaine Hydrochloride
  Arms: Clo-TAP (Bupi + Clon); TAP (Bupi)
Drug: Clonidine — 2 x 1ml Clonidine = 150 µg Clonidine
  Other Names: Clonidine Hydrochloride
  Arms: Clo-TAP (Bupi + Clon)

SUMMARY:
The purpose of this study is to determine whether a transversus abdominis plane (TAP) block with Clonidine added to the injectate (Clo-TAP) performed approximately 2hrs after the cesarean section (CS) will decrease the amount of postoperative hyperalgesia and ultimately reduce post-CS chronic pain.

DETAILED DESCRIPTION:
Acute severe pain after cesarean section (CS) occurs more often than is thought and 10-15% of the women having a cesarean section develop chronic pain (Kehlet et al. 2006). With over 1.3 million cesarean deliveries per year in the US, this is bound to create a significant health problem. One way to address this health burden is to refine techniques that may help control the pain women experience after CS and ultimately reduce the potential to develop chronic pain.

The purpose of this randomized, double-blinded study is to evaluate the ability of an established anesthetic technique called the transversus abdominis plane (TAP) block to reduce the amount of hyperalgesia women develop around their incision after CS. Measuring the amount of punctuate mechanical hyperalgesia is used as a tool to assess postoperative central sensitization (Lavand'homme et al. 2005), which contributes to postoperative acute pain. Since postoperative acute pain has been shown to be predictive of developing postoperative chronic pain (Eisenach et al. 2008; Yarnitsky et al. 2008), an effective TAP block could help diminish the incidence of chronic pain after CS. In addition, blood samples will be collected for future genetic analysis and we will test preoperatively for mechanical temporal summation (mTS) to evaluate CNS (central nervous system) sensitization and nociceptive system hyperexcitability and see if this correlates with the amount of hyperalgesia women develop around their incision after surgery.

The primary aim of this study is to evaluate the benefits of two different solutions injected by TAP block technique on postoperative peri-incisional hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* non-laboring women who will benefit from and have clinically consented to a scheduled or non-scheduled cesarean delivery under spinal anesthesia
* English speaking (UW Site) or Portuguese speaking (Brazil site)
* aged between 18 and 45 years
* BMI < 40
* ASA physical status class I or II

Exclusion Criteria:

* laboring women undergoing a non-scheduled cesarean delivery
* non-English speaking (UW Site) or non-Portuguese speaking (Brazil site)
* previous spinal surgery
* contraindications for neuraxial anesthesia
* allergy to local anesthetic, ultrasound conduction gel, or Clonidine
* history of chronic pain
* inability to receive intraoperative Toradol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Landau, MD, Study Chair — University of Washington; Laurent Bollag, MD, Principal Investigator — University of Washington
Locations (2):
- University of Washington, Seattle, Washington, United States
- Hospital e Maternidade Santa Joana, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchanan ML, Easterling TR, Carr DB, Shen DD, Risler LJ, Nelson WL, Mattison DR, Hebert MF. Clonidine pharmacokinetics in pregnancy. Drug Metab Dispos. 2009 Apr;37(4):702-5. doi: 10.1124/dmd.108.024984. Epub 2008 Dec 30. PMID 19116263
- [Background] Carvalho B, Angst MS, Fuller AJ, Lin E, Mathusamy AD, Riley ET. Experimental heat pain for detecting pregnancy-induced analgesia in humans. Anesth Analg. 2006 Nov;103(5):1283-7. doi: 10.1213/01.ane.0000239224.48719.28. PMID 17056970
- [Background] Duma A, Urbanek B, Sitzwohl C, Kreiger A, Zimpfer M, Kapral S. Clonidine as an adjuvant to local anaesthetic axillary brachial plexus block: a randomized, controlled study. Br J Anaesth. 2005 Jan;94(1):112-6. doi: 10.1093/bja/aei009. Epub 2004 Oct 29. PMID 15516351
- [Background] Eisenach JC, De Kock M, Klimscha W. alpha(2)-adrenergic agonists for regional anesthesia. A clinical review of clonidine (1984-1995). Anesthesiology. 1996 Sep;85(3):655-74. doi: 10.1097/00000542-199609000-00026. No abstract available. PMID 8853097
- [Background] Gabriel JS, Gordin V. Alpha 2 agonists in regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2001 Dec;14(6):751-3. doi: 10.1097/00001503-200112000-00024. PMID 17019175
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Landau R, Schiffer E, Morales M, Savoldelli G, Kern C. The dose-sparing effect of clonidine added to ropivacaine for labor epidural analgesia. Anesth Analg. 2002 Sep;95(3):728-34, table of contents. doi: 10.1097/00000539-200209000-00036. PMID 12198061
- [Background] Lavand'homme P. Postcesarean analgesia: effective strategies and association with chronic pain. Curr Opin Anaesthesiol. 2006 Jun;19(3):244-8. doi: 10.1097/01.aco.0000192815.22989.61. PMID 16735805
- [Background] Lavand'homme P. Perioperative pain. Curr Opin Anaesthesiol. 2006 Oct;19(5):556-61. doi: 10.1097/01.aco.0000245284.53152.1f. PMID 16960491
- [Background] Lavand'homme P, De Kock M, Waterloos H. Intraoperative epidural analgesia combined with ketamine provides effective preventive analgesia in patients undergoing major digestive surgery. Anesthesiology. 2005 Oct;103(4):813-20. doi: 10.1097/00000542-200510000-00020. PMID 16192774
- [Background] Lavand'homme PM, Roelants F, Waterloos H, Collet V, De Kock MF. An evaluation of the postoperative antihyperalgesic and analgesic effects of intrathecal clonidine administered during elective cesarean delivery. Anesth Analg. 2008 Sep;107(3):948-55. doi: 10.1213/ane.0b013e31817f1595. PMID 18713912
- [Background] Lavand'homme PM, Roelants F, Waterloos H, De Kock MF. Postoperative analgesic effects of continuous wound infiltration with diclofenac after elective cesarean delivery. Anesthesiology. 2007 Jun;106(6):1220-5. doi: 10.1097/01.anes.0000267606.17387.1d. PMID 17525598
- [Background] Marhofer P, Greher M, Kapral S. Ultrasound guidance in regional anaesthesia. Br J Anaesth. 2005 Jan;94(1):7-17. doi: 10.1093/bja/aei002. Epub 2004 Jul 26. PMID 15277302
- [Background] McCartney CJ, Duggan E, Apatu E. Should we add clonidine to local anesthetic for peripheral nerve blockade? A qualitative systematic review of the literature. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):330-8. doi: 10.1016/j.rapm.2007.02.010. PMID 17720118
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] McDonnell JG, Laffey JG. Transversus abdominis plane block. Anesth Analg. 2007 Sep;105(3):883. doi: 10.1213/01.ane.0000268542.45107.79. No abstract available. PMID 17717264
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] Mendez R, Eisenach JC, Kashtan K. Epidural clonidine analgesia after cesarean section. Anesthesiology. 1990 Nov;73(5):848-52. doi: 10.1097/00000542-199011000-00009. PMID 2240674
- [Background] Nikolajsen L, Sorensen HC, Jensen TS, Kehlet H. Chronic pain following Caesarean section. Acta Anaesthesiol Scand. 2004 Jan;48(1):111-6. doi: 10.1111/j.1399-6576.2004.00271.x. PMID 14674981
- [Background] Ohel I, Walfisch A, Shitenberg D, Sheiner E, Hallak M. A rise in pain threshold during labor: a prospective clinical trial. Pain. 2007 Nov;132 Suppl 1:S104-S108. doi: 10.1016/j.pain.2007.05.007. Epub 2007 Jun 20. PMID 17583429
- [Background] Pan PH, Coghill R, Houle TT, Seid MH, Lindel WM, Parker RL, Washburn SA, Harris L, Eisenach JC. Multifactorial preoperative predictors for postcesarean section pain and analgesic requirement. Anesthesiology. 2006 Mar;104(3):417-25. doi: 10.1097/00000542-200603000-00007. PMID 16508387
- [Background] Parker RK, Connelly NR, Lucas T, Serban S, Pristas R, Berman E, Gibson C. Epidural clonidine added to a bupivacaine infusion increases analgesic duration in labor without adverse maternal or fetal effects. J Anesth. 2007;21(2):142-7. doi: 10.1007/s00540-006-0476-8. Epub 2007 May 30. PMID 17458641
- [Background] Weissman-Fogel I, Granovsky Y, Crispel Y, Ben-Nun A, Best LA, Yarnitsky D, Granot M. Enhanced presurgical pain temporal summation response predicts post-thoracotomy pain intensity during the acute postoperative phase. J Pain. 2009 Jun;10(6):628-36. doi: 10.1016/j.jpain.2008.12.009. Epub 2009 Apr 23. PMID 19398382
- [Background] Yarnitsky D, Crispel Y, Eisenberg E, Granovsky Y, Ben-Nun A, Sprecher E, Best LA, Granot M. Prediction of chronic post-operative pain: pre-operative DNIC testing identifies patients at risk. Pain. 2008 Aug 15;138(1):22-28. doi: 10.1016/j.pain.2007.10.033. Epub 2008 Jan 8. PMID 18079062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | TAP (Bupi) | Clo-TAP (Bupi + Clon)
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAP (Bupi) | Clo-TAP (Bupi + Clon) | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.7) | 31.8 (4.5) | 29.5 (6.7) | 30 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 30 | 90
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Wound Hyperalgesia Index (WHA) Assessed 48 Hrs After Block Placement in the Different Groups
Description: Determine which of three different TAP formulations (Placebo, TAP, Clo-TAP) has the most beneficial effect on the postoperative area of hyperalgesia 48hrs after the start of the cesarean section. The smaller the area of WHA, assessed in cm2, the better the outcome. Area sizes may range from 0 to any size.
Time Frame: 48hrs after CS
Measure: Mean (Inter-Quartile Range); unit: cm^2
Arm/Group | Placebo | TAP (Bupi) | Clo-TAP (Bupi + Clon)
Number analyzed (Participants) | 30 | 30 | 30
cm^2 | 1.07 [0.48 to 3.26] | 1.27 [0.59 to 2.95] | 0.74 [0.09 to 2.25]
Statistical Analysis 1: Comparison: Placebo vs TAP (Bupi) vs Clo-TAP (Bupi + Clon); We estimated that 25 subjects per group would allow us to detect a reduction of this area from 7.5 cm2 in our placebo group to 3.5 cm2 in the CloTAP group, with SD = 5 cm2 in both groups, owing to improved overall analgesia and reduced pain sensitization in women allocated to receive a TAP block with clonidine (2-tailed [alpha] = 0.05, 80% power). To allow for failed TAP blocks and/or exclusions of cases, we included 30 patients per group (n = 90); Test type: Other; p = 0.48, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo | TAP (Bupi) | Clo-TAP (Bupi + Clon)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | TAP (Bupi) (N=30) | Clo-TAP (Bupi + Clon) (N=30)
LAST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — Local anesthetic systemic toxicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes